CLINICAL TRIAL: NCT00001971
Title: Evaluation of Patients With Liver Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910214; 91-DK-0214
Record Dates: First submitted 2006-07-12; First posted 2000-01-19 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-30

CONDITIONS: Hepatitis D; Hepatitis C; Hepatitis B; Liver Disease
Keywords: Hepatitis B; Hepatitis C; Hepatitis D; Chronic Hepatitis; Natural History; Liver Disease
MeSH Terms: conditions — Hepatitis D; Hepatitis C; Hepatitis B; Liver Diseases; Hepatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy individuals: Healthy individuals who have recovered from liver diseases or who are healthy volunteers
- Patients: Liver disease patients

SUMMARY:
The proposed study aims to evaluate, investigate, and follow-up patients suffering from acute and chronic liver disease. The study will focus on understanding diseases affecting the liver.

Patients participating in the study will first undergo a routine check-up as an outpatient. They will be asked to provide blood and urine samples for laboratory testing and will undergo an ultrasound of the liver. Ultrasound examinations use sound waves to determine the size and texture of the liver. After the initial visit subjects will be requested to follow-up once a year at the outpatient department for a similar check-up.

Additional tests may be requested throughout the study to provide information for other research studies and individual consent will be requested. These tests may include liver biopsies, skin biopsies, and / or specialized blood, plasma, and lymphocyte examinations.

Subjects that qualify for medications presently being studied may be offered the opportunity to benefit from experimental therapy.

DETAILED DESCRIPTION:
Study Description:

This is a clinical research protocol to allow for collection of samples and data obtained during clinical evaluation and long-term follow up of patients who have an acute or chronic liver disease. The protocol is designed to create a repository to study the natural history and pathogenesis of various liver diseases such as acute and chronic hepatitis B, C, D and E, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, hemochromatosis, nonalcoholic steatohepatitis (NASH), noncirrhotic portal hypertension, hepatocellular carcinoma, and cryptogenic or poorly defined forms of chronic liver disease. Samples collected during the course of clinical care for patients with liver disease include blood, saliva, urine, stool, and residual tissue obtained during clinically-indicated liver biopsies not otherwise needed for clinical care. Additionally, subjects with liver disease will be asked to provide a blood sample for genetic analysis. Healthy volunteers will be recruited and asked to provide a blood sample to serve as controls for the genetic analyses. Research will be conducted to investigate genetic factors that may contribute to liver diseases

Objectives: Primary Objective

To collect data and samples during clinical evaluation, treatment and follow-up of participants for future use in studies of liver diseases

Secondary Objective

To determine if genetic factors may contribute to the susceptibility, progression, outcome, or treatment success of different liver diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected Subjects

In order to be eligible to participate in this study, an affected participant must meet all of the following criteria:

1. >=2 years of age.
2. Meets one of the following:

   1. Suspected or evidence of acute or chronic liver disease on evaluation by a referring licensed independent practitioner (LIP), OR
   2. At risk for acute or chronic liver disease

Healthy Volunteers

In order to be eligible to participate in this study, a healthy volunteer must meet all of the following criteria:

1. >= 18 years of age.
2. In good general health as evidenced by medical history

EXCLUSION CRITERIA:

Affected Participants

An affected participant who meets any of the following criteria will be excluded from participation in this study:

1. History of significant medical illnesses that might interfere with prolonged follow up evaluation

Healthy Volunteers

A healthy volunteer who meets any of the following criteria will be excluded from participation in this study:

1. Any chronic medical condition, including (but not limited to) heart, kidney, or lung diseases
2. Taking any regular medications or supplements (with the exception of regular multivitamins and/or oral contraceptives)
3. Average alcohol consumption > 1 drink/day in past 6 months, per self-report
4. History of liver disease (with the exception of neonatal jaundice)
5. History of severe illness, infection or major surgery in the past year
6. History of cancer (with the exception of basal cell carcinoma resected > 1 year prior to enrollment)
7. BMI < 18 or BMI >25
8. Hemoglobin < 11 (women) or hemoglobin < 12 (men)
9. ALT >35 (men) or ALT >25 (women)
10. Alkaline Phosphatase >= 150
11. Bilirubin >2 g/dL
12. HIV positive, Anti-HCV positive, HBsAg positive or Anti-HBc positive
13. Pregnancy
14. Inability to provide informed consent

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a general clinical research protocol to allow for evaluation, investigation and long-term follow up of patients who have an acute or chronic liver disease. The protocol is designed to study the natural history and pathogenesis of various liver diseases such as acute and chronic hepatitis B, C, D and E, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, hemochromatosis, nonalcoholic steatohepatitis (NASH), noncirrhotic portal hypertension, hepatocellular carcinoma, and cryptogenic or poorly defined forms of chronic liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 8050 (Estimated)
Dates: Start 1992-05-27 (Actual)

PRIMARY OUTCOMES:
Predisposition and outcomes related to liver disease susceptibility, progression, and treatment response | Annual visits
  Predisposition and outcomes related to liver disease susceptibility, progression, and treatment response

CONTACTS AND LOCATIONS:
Overall Officials: T. Jake Liang, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali RO, Moon MS, Townsend EC, Hill K, Zhang GY, Bradshaw A, Guan H, Hamilton D, Kleiner DE, Auh S, Koh C, Heller T. Exploring the Link Between Platelet Numbers and Vascular Homeostasis Across Early and Late Stages of Fibrosis in Hepatitis C. Dig Dis Sci. 2020 Feb;65(2):524-533. doi: 10.1007/s10620-019-05760-x. Epub 2019 Aug 12. PMID 31407130
- [Derived] Kefalakes H, Koh C, Sidney J, Amanakis G, Sette A, Heller T, Rehermann B. Hepatitis D Virus-Specific CD8+ T Cells Have a Memory-Like Phenotype Associated With Viral Immune Escape in Patients With Chronic Hepatitis D Virus Infection. Gastroenterology. 2019 May;156(6):1805-1819.e9. doi: 10.1053/j.gastro.2019.01.035. Epub 2019 Jan 18. PMID 30664876
- [Derived] Koh C, Turner T, Zhao X, Minniti CP, Feld JJ, Simpson J, Demino M, Conrey AK, Jackson MJ, Seamon C, Kleiner DE, Kato GJ, Heller T. Liver stiffness increases acutely during sickle cell vaso-occlusive crisis. Am J Hematol. 2013 Nov;88(11):E250-4. doi: 10.1002/ajh.23532. Epub 2013 Aug 1. PMID 23828202
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1991-DK-0214.html